CLINICAL TRIAL: NCT02220361
Title: Phase 4 Study of Effects of Dexmedetomidine on Prevention of Side Effects of Hemabate in Cesarean Section Patients
Brief Title: Dexmedetomidine on Prevention of Side Effects of Hemabate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jin Ni (Other)
Responsible Party: Sponsor-Investigator, Jin Ni, Department of Anesthesiology, Guangzhou Women and Children's Medical Center
Organization: Guangzhou Women and Children's Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JNi; DAGZWCMC (Other: Department of Anesthesiology,Guangzhou Women and Children's Medical Center)
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Gynecological Patient
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo group (Placebo Comparator): received 20 ml intravenous physiological saline
  Interventions: Drug: placebo
- low dose dexmedetomidine group (Experimental): received 0.5μgkg-1 intravenous dexmedetomidine (Jiang Su Heng Rui Medicine Co. Ltd, Jiangsu Province, China) diluted to 20ml with physiological saline
  Interventions: Drug: low dose dexmedetomidine
- hemabate+high dose dexmedetomidine group (Experimental): received 1μgkg-1 intravenous dexmedetomidine (Jiang Su Heng Rui Medicine Co. Ltd, Jiangsu Province, China) diluted to 20ml with physiological saline
  Interventions: Drug: high dose dexmedetomidine

INTERVENTIONS:
Drug: placebo — received 20 ml intravenous physiological saline The infusion were completed in 30 minutes.
  Arms: placebo group
Drug: low dose dexmedetomidine — received 0.5μgkg-1 intravenous dexmedetomidine (Jiang Su Heng Rui Medicine Co. Ltd, Jiangsu Province, China) diluted to 20ml with physiological saline The infusion were completed in 30 minutes.
  Arms: low dose dexmedetomidine group
Drug: high dose dexmedetomidine — received 1μgkg-1 intravenous dexmedetomidine (Jiang Su Heng Rui Medicine Co. Ltd, Jiangsu Province, China) diluted to 20ml with physiological saline.
  The infusion was completed in 30 minutes
  Arms: hemabate+high dose dexmedetomidine group

SUMMARY:
Hemabate is often used for gynecological patients. Hemabate is associated with many side effects, including a burning sensation in the stomach, nausea, vomiting, diarrhea etc. It is reported that dexmedetomidine reduce gastrointestinal reaction during perioperative period. We design this clinical trial to find if dexmedetomidine can prevent the side effects of hemabate in Cesarean Section patients.

ELIGIBILITY:
Inclusion Criteria:

gynecological patients

Exclusion Criteria:

* Neuromuscular and endocrine diseases
* Allergic reactions to a2-adrenergic agonist
* Previous abdominal surgery including prior caesarean section.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
SpO2 Change | participants will be followed for the duration of surgery, an expected average of 2 hours
systolic blood pressure and diastolic blood pressure change | participants will be followed for the duration of surgery, an expected average of 2 hours
Heart rate change | participants will be followed for the duration of surgery, an expected average of 2 hours
nausea | 24 h postoperatively
vomiting | 24h postoperatively
fever | 24h postoperatively
diarrhea | 24h postoperatively
headache | 24h postoperatively
elevated blood pressure | 24h postoperatively
chest congestion | 24h postoperatively